CLINICAL TRIAL: NCT06159036
Title: Effects of a Strength Training Program in Inertial Machines on Squat Jump, Countermovement Jump and Abalakov in Youth Volleyball Players
Brief Title: Effects of a Strength Training Program in Inertial Machines on Bosco Test in Youth Volleyball Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Autónoma de Manizales, Colombia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: APPROVAL ACT 07-19-2022_11UAM
Record Dates: First submitted 2023-02-03; First posted 2023-12-06 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-12

CONDITIONS: Volleyball; Player; Female
Keywords: Keywords: Inertial machines; Squat jump; Countermovent Jump; Abalakov

STUDY DESIGN:
Intervention Model Description: The athletes were divided into two experimental and control groups, for which the experimental group was asked to carry out a protocol that consisted of 12 weeks of intervention divided in a randomized manner, resulting in a pre and post intervention measurement
Who Masked: Investigator
Masking Description: One of the main researchers evaluated the post-test without knowing who belonged to the control and experimental group, in addition to this, the other investigator was asked to evaluate the pre-test so as not to have biases or generate some type of modification in the results obtained by both groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Strength training in inertial machines for 2 days and around 12 weeks.
  Interventions: Device: Inertial Strength training
- Group 2 (Active Comparator): Control group developed conventional strength training with squats, deadlifts, hip thrust jumps for 2 days and around 12 weeks.
  Interventions: Device: Inertial Strength training

INTERVENTIONS:
Device: Inertial Strength training — Low speed strength training with classic movements, derived from Olympic lifting and jumping
  Other Names: Conventional strength training

SUMMARY:
Objective: To determine the effect of strength training in inertial machines, on SJ CMJ and CMJ with arms; in youth volleyball players from the city of Cartago.

Methodology: A quasi-experimental study of quantitative order was carried out and takes up an empirical-analytical approach, quasi-experimental with pre-test - post-test evaluation. 32 female volleyball players, belonging to the minor category of the Fénix G Club of the city of Cartago Valle

Results: Both groups showed significant improvements in jump height, flight time, strength and power in the protocol that was carried out during the 12 weeks of intervention, but there was no statistically significant difference between the control groups (P = 0.356). , experimental (P = 0.984)

Conclusions:

Keywords: Inertial machines, Squat jump, Countermovent Jump, Abalakov

DETAILED DESCRIPTION:
Objective: To determine the effect of strength training in inertial machines, on SJ CMJ and CMJ with arms; in youth volleyball players from the city of Cartago.

Methodology: A quasi-experimental study of quantitative order was carried out and takes up an empirical-analytical approach, quasi-experimental with pre-test - post-test evaluation. 32 female volleyball players, belonging to the minor category of the Fénix G Club of the city of Cartago Valle. The techniques that were used were: survey to determine previous injuries, adaptations that athletes may have against strength training and practice time in volleyball, observations were also developed to determine the levels of jumpability of each player, taking into account the Bosco's battery (3). For this we used:

* My jumps 2 application for IOS devices, it was used to determine the height of the CMJ, SJ, CMJ or ABK, this app was validated in 2015 by the creator, Dr. Carlos Balsalobre (15).
* Wheeler YOYO XS inertial machine contains an encoder validated by the company Chronjump (16) with this device the training program was carried out with the volleyball players, the program was subjected to expert judgment.

For the collection of information on sociodemographic variables, a data record was carried out (Weight, Height, History of injuries, etc.), in addition to this, a record per athlete for the values of each jump performed.

Results: Both groups showed significant improvements in jump height, flight time, strength and power in the protocol that was carried out during the 12 weeks of intervention, but there was no statistically significant difference between the control groups (P = 0.356). , experimental (P = 0.984)

Conclusions:

Keywords: Inertial machines, Squat jump, Countermovent Jump, Abalakov

ELIGIBILITY:
Inclusion criterio

* That they express their participation voluntarily in the investigation by filling out their informed consent in the informed settlement.
* Sports aptitude in the execution of the tests at the time of the intervention and/or evaluation, do not present any surgical intervention in any particular area or region of the lower limbs.
* Practice time in volleyball of at least 2 years and 1 year in strength training

Exclusion Criteria:

* Presenting serious sports injuries 6 months before or during the data collection phase (pre-test and post-test) and application of training with inertial machines.
* not complete with at least 8 weeks of strength training on the inertial machine.

Ages: 15 Years to 17 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — According to the availability of the subjects.
Enrollment: 30 (Actual)
Dates: Start 2022-09-26 (Actual); Primary Completion 2022-11-24 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Independent variable: Inertial machine program | 12 weeks of intervention
  Power (watt)
Dependent variable: countermovement jump, squat jump and abalakov. | 12 weeks of intervention
  Squat position with arms at the waist looking for a countermovement and height, the following jump squat position hold for 5 seconds and look for height without taking the hands off the waist, finally the abalakov is a jump with loose arms performing a countermovement and looking height.

SECONDARY OUTCOMES:
To compare the differences pre and post strength training in inertial versus conventional machines, pre-post control experiment on the SJ, CMJ and ABK in youth volleyball players. | 12 weeks of intervention
  Squat position with arms at the waist looking for a countermovement and height, the following jump squat position hold for 5 seconds and look for height without taking the hands off the waist, finally the abalakov is a jump with loose arms performing a countermovement and looking height.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Autónoma de Manizales, Manizales, Caldas Department, Colombia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Balsalobre-Fernandez C, Glaister M, Lockey RA. The validity and reliability of an iPhone app for measuring vertical jump performance. J Sports Sci. 2015;33(15):1574-9. doi: 10.1080/02640414.2014.996184. Epub 2015 Jan 2. PMID 25555023
- [Result] Penailillo L, Blazevich A, Numazawa H, Nosaka K. Metabolic and muscle damage profiles of concentric versus repeated eccentric cycling. Med Sci Sports Exerc. 2013 Sep;45(9):1773-81. doi: 10.1249/MSS.0b013e31828f8a73. PMID 23475167
- [Result] Beato M, Dello Iacono A. Implementing Flywheel (Isoinertial) Exercise in Strength Training: Current Evidence, Practical Recommendations, and Future Directions. Front Physiol. 2020 Jun 3;11:569. doi: 10.3389/fphys.2020.00569. eCollection 2020. No abstract available. PMID 32581845
- [Result] Martinez-Aranda LM, Fernandez-Gonzalo R. Effects of Inertial Setting on Power, Force, Work, and Eccentric Overload During Flywheel Resistance Exercise in Women and Men. J Strength Cond Res. 2017 Jun;31(6):1653-1661. doi: 10.1519/JSC.0000000000001635. PMID 28538317